CLINICAL TRIAL: NCT02698800
Title: Blocking Nocturnal Blue Light to Treat Insomnia: A Pilot Randomized Controlled Trial
Brief Title: Blue Blockers at Night and Insomnia Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Ari Shechter, Assistant Professor of Medical Sciences (in Medicine), Columbia University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AAAQ6404
Record Dates: First submitted 2016-02-26; First posted 2016-03-04 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Insomnia; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Lenses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blue blocking (BB) (Experimental): Wearing of BB lenses.
  Interventions: Device: Blue blocking (BB) lenses
- Clear (Placebo Comparator): Wearing of clear lenses
  Interventions: Device: Clear lenses

INTERVENTIONS:
Device: Blue blocking (BB) lenses — Participants will wear blue blocking lenses each night for 1 week for 2 hours preceding bedtime.
  Arms: Blue blocking (BB)
Device: Clear lenses — Participants will wear clear lenses each night for 1 week for 2 hours preceding bedtime.
  Arms: Clear

SUMMARY:
Under entrained conditions, humans maintain a consolidated nocturnal sleep episode that coincides with environmental darkness and endogenous melatonin secretion. Various factors, such as artificial light, can compromise this temporal harmony, resulting in sleep disruption. Light is the strongest synchronizer of the circadian clock, with direct inputs via the retinohypothalamic tract to brain centers regulating sleep and circadian rhythms. Evening light exposure can suppress melatonin secretion and worsen sleep. This is critical, since most individuals routinely expose themselves to light before bedtime. The high sensitivity of the circadian system to blue wavelength light indicates that modern light sources such as light-emitting diodes (LED) may have particularly deleterious effects on sleep. It is possible to selectively filter out blue light while maintaining other visible spectra with blue-blocking (BB) lenses. Wearing BB lenses before bedtime may present a simple, affordable, and safe method to improve sleep. None have yet investigated the effects of BB lenses on subjective and objective sleep in insomnia patients, while simultaneously exploring the effects on melatonin secretion.

DETAILED DESCRIPTION:
This study seeks to investigate the impact of BB lenses on melatonin and sleep in insomnia patients using a randomized, placebo-controlled crossover study, with the aim of developing a novel non-pharmacological approach for the treatment of insomnia. 15 individuals with insomnia will wear either BB or placebo (clear) lenses for 2 hours preceding bedtime while at home, for 1 week in a cross-over design. Sleep quality will be documented while at home, at also melatonin secretion while in the laboratory. It is predicted that compared to placebo, wearing BB lenses for 2 hours preceding bedtime will attenuate bright light associated melatonin suppression and improve sleep.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia for at least 1 month based on Insomnia Symptoms Questionnaire

Exclusion Criteria:

* obstructive sleep apnea; narcolepsy; periodic leg movement disorder
* currently shift worker
* psychiatric or neurologic disorders
* deep vein thrombosis
* current cigarette smoker
* currently taking beta-blockers
* pregnant/breastfeeding
* children less than 1 year old at home
* excessive daily caffeine intake

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari Shechter, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shechter A, Kim EW, St-Onge MP, Westwood AJ. Blocking nocturnal blue light for insomnia: A randomized controlled trial. J Psychiatr Res. 2018 Jan;96:196-202. doi: 10.1016/j.jpsychires.2017.10.015. Epub 2017 Oct 21. PMID 29101797
- [Derived] Shechter A, Westwood AJ. A behavioral intervention for insomnia improves blood pressure. Sleep Med. 2017 Sep;37:225. doi: 10.1016/j.sleep.2017.07.003. Epub 2017 Jul 15. No abstract available. PMID 28760541

RESULTS

PARTICIPANT FLOW:
Groups:
- BB First (7 d), Then Clear (7 d), Separated by 4-wk Washout: Wearing of BB first for 7 days, followed by Clear lenses for 7 days, separated by 4-week washout period
  Blue blocking (BB) lenses: Participants will wear blue blocking lenses each night for 1 week for 2 hours preceding bedtime.
  Clear lenses: Participants will wear clear lenses each night for 1 week for 2 hours preceding bedtime
- Clear First (7 ), Then BB (7 d), Separated by 4-wk Washout: Wearing Clear lenses first for 7 days, followed by BB lenses for 7 days, separated by a 4-week washout period
Period: Overall Study
Arm/Group | BB First (7 d), Then Clear (7 d), Separated by 4-wk Washout | Clear First (7 ), Then BB (7 d), Separated by 4-wk Washout
Started | 7 | 8
Completed | 6 | 8
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Individuals with insomnia symptoms
Groups:
- Blue Blocking (BB)/Clear: Wearing of BB lenses.
  Blue blocking (BB) lenses: Participants will wear blue blocking lenses each night for 1 week for 2 hours preceding bedtime.
  Clear lenses: Participants will wear clear lenses each night for 1 week for 2 hours preceding bedtime.
Arm/Group | Blue Blocking (BB)/Clear
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black/African American | 6
  White | 6
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Pittsburgh Insomnia Rating Scale-65 (PIRS65) Total Score
Description: Pittsburgh Insomnia Rating Scale-65; measures the self-reported severity of insomnia over the past week. Higher scores indicate worsened severity. There are 65 items, each scored on a 4-point scale from low-high on symptom severity or frequency. There is a Total score, and 3 subscales: Distress score (how bothersome the sleep impairment is), Sleep Parameters score (sleep quality), and Quality of Life score.
  For the total score scoring is done by summing the scores from questions 1-65. Minimum Score=0 (good); Maximum Score=195 (bad) For the distress score, scoring is done by summing the scores from questions 1-46. Minimum Score=0 (not bothered); Maximum Score=138 (severely bothered) For the sleep parameters score, scoring is done by summing the scores from questions 47-56. Minimum Score=0 (good sleep); Maximum Score=30 (disrupted sleep) For the quality of life score, scoring is done by summing the scores from questions 57-65. Minimum Score=0 (excellent); Maximum Score=27 (poor)
Time Frame: After 7 nights of BB lenses
Population: Participants who completed both phases
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blue Blocking (BB)
Number analyzed (Participants) | 14
units on a scale | 72.64 (28.14)

2. Primary Outcome: Pittsburgh Insomnia Rating Scale-65 (PIRS65) Total Score
Description: as for outcome 1
Time Frame: After 7 nights of clear lenses
Population: Participants who complete both phases
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clear
Number analyzed (Participants) | 14
units on a scale | 88.93 (33.19)

3. Secondary Outcome: Sleep Efficiency (Time Spent Asleep Divided by Total Time in Bed) Determined With Wrist-worn Accelerometry
Description: Wrist-worn accelerometry gives an estimate of time spent asleep, time spent in bed, and sleep efficiency can be calculated from this. Sleep efficiency is calculated as time spent asleep divided by total time in bed. Here, we considered the mean calculated sleep efficiency over each 7-day treatment period.
Time Frame: After 7 nights of BB lenses
Population: Participants who completed both phases
Measure: Mean (Standard Deviation); unit: % of total sleep time
Arm/Group | Blue Blocking (BB)
Number analyzed (Participants) | 14
% of total sleep time | 78.35 (9)

4. Secondary Outcome: Sleep Efficiency (Time Spent Asleep Divided by Total Time in Bed) Determined With Wrist-worn Accelerometry
Description: as for outcome 3
Time Frame: After 7 nights of clear lenses
Population: Participants who completed both phases
Measure: Mean (Standard Deviation); unit: % of total sleep time
Arm/Group | Clear
Number analyzed (Participants) | 14
% of total sleep time | 77.01 (8.67)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: This was a minimal risk intervention, with no expected adverse events
Arm/Group | Blue Blocking (BB) | Clear
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT02698800/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT02698800/ICF_001.pdf